CLINICAL TRIAL: NCT00318292
Title: Preemptive Local Anesthesia in Vaginal Surgery, A Prospective, Randomised Trial
Brief Title: Preemptive Local Anesthesia in Vaginal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Jeffrey Cornella MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 63-06
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Results first posted 2009-03-18 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-10

CONDITIONS: Pain, Postoperative
Keywords: preemptive analgesia; paracervical block; vaginal hysterectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PLA (Experimental): Active preemptive local analgesia.
  Interventions: Drug: bupivacaine and epinephrine
- Placebo (Placebo Comparator): Placebo for preemptive local analgesia.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: bupivacaine and epinephrine — 20 ml of 0.5% bupivacaine with 1:200,000 epinephrine paracervical injection.
  Arms: PLA
Drug: Placebo — 20 ml normal saline injection.
  Arms: Placebo

SUMMARY:
Preemptive analgesia is an intervention which provides an anesthetic prior to initiating a painful stimulus. This trial is examining the effects of a local anesthetic given at the point of innervation prior to performing a vaginal hysterectomy with suspension sutures.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing vaginal hysterectomy with McCall's culdoplasty

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime B. Long, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States

REFERENCES:
- [Result] Long JB, Eiland RJ, Hentz JG, Mergens PA, Magtibay PM, Kho RM, Magrina JF, Cornella JL. Randomized trial of preemptive local analgesia in vaginal surgery. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Jan;20(1):5-10. doi: 10.1007/s00192-008-0716-6. Epub 2008 Oct 2. PMID 18830553

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing vaginal hysterectomy with McCall culdoplasty at the Mayo Clinic Hospital were recruited from 17 May 2006 to 14 February 2008. We screened 146 patients who were scheduled for vaginal surgery, and 142 were eligible to participate.
Pre-assignment Details: 95 of the eligible patients consented to participate. 3 were excluded prior to treatment because they converted to abdominal hysterectomy. 2 were excluded because the study treatment was unintentionally missed by the operating staff.
Groups:
- Preemptive Local Analgesia (PLA): Active preemptive local analgesia.
Period: Overall Study
Arm/Group | Preemptive Local Analgesia (PLA) | Placebo
Started | 45 | 45
Completed | 45 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preemptive Local Analgesia (PLA) | Placebo | Total
Number analyzed (Participants) | 45 | 45 | 90
Age Continuous [Mean (Standard Deviation); unit: years] | 57 (15) | 54 (20) | 56 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 90
  Male | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 26.2 (5.4) | 25.4 (4.0) | 25.8 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS) Pain Score
Description: Visual Analogue Scale (VAS) pain score on a scale from 0 (None) to 10 (Worst) points.
Time Frame: 30 minutes post-op
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Preemptive Local Analgesia (PLA) | Placebo
Number analyzed (Participants) | 45 | 45
points on a scale | 2.5 (3.1) | 4.4 (3.0)
Statistical Analysis 1: Comparison: Preemptive Local Analgesia (PLA) vs Placebo; Test type: Superiority or Other; p = .003, t-test, 2 sided; Mean Difference (Final Values) = -1.9, 95% CI [-3.2 to -0.7]

ADVERSE EVENTS:
Time Frame: 6 weeks.
Arm/Group | Preemptive Local Analgesia (PLA) | Placebo
Serious Adverse Events (participants affected / at risk) | 5/45 | 3/45
Other Adverse Events (participants affected / at risk) | 18/45 | 22/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preemptive Local Analgesia (PLA) (N=45) | Placebo (N=45)
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Bacterial Infection (Infections and infestations) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postoperative Nausea and Vomiting Requiring Readmission (Gastrointestinal disorders) | 0 | 1
Postoperative Pain Requiring Readmission (Surgical and medical procedures) | 2 | 0
Pulmonary Embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preemptive Local Analgesia (PLA) (N=45) | Placebo (N=45)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rectal Pain (Surgical and medical procedures) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 16 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes